CLINICAL TRIAL: NCT07334795
Title: Intermountain Stewardship in Community Outpatient Settings-Resources & Engagement-Pediatrics
Acronym: SCORE-Peds
Status: Not yet recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: HSII_IHC_IMP-PS2
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Infection (for Example, Pneumonia, Bronchitis); Antibiotic; Antibiotic Duration; Antibiotic Prescribing for Acute Respiratory-tract Infections
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia; Bronchitis | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with ARTIs, Wave 1: Children under 18 treated in Wave 1 of antibiotic stewardship for the following conditions: acute otitis media (AOM), Group A Streptococcal (GAS) pharyngitis, acute sinusitis, and community-acquired pneumonia (CAP)
  Interventions: Other: Implementation strategies including training & education, EMR tools, audit & feedback reports, and facilitation
- Children with ARTIs, Wave 2: Children under 18 treated in Wave 2 of antibiotic stewardship for the following conditions: acute otitis media (AOM), Group A Streptococcal (GAS) pharyngitis, acute sinusitis, and community-acquired pneumonia (CAP)
  Interventions: Other: Implementation strategies including training & education, EMR tools, audit & feedback reports, and facilitation

INTERVENTIONS:
Other: Implementation strategies including training & education, EMR tools, audit & feedback reports, and facilitation — o facilitate improved adherence to guideline-based prescribing, we plan a variety of implementation strategies to be employed in tandem including training & education, EMR tools (e.g., Smart sets, express lanes, preference lists), audit and feedback reports and dashboards, and facilitation.

SUMMARY:
The goal of this implementation project is to detail the process of implementing the best practice of antibiotic stewardship in the pediatric population across the Intermountain Health medical system. The main questions it aims to answer are:

* How can a large healthcare system drive high adherence to antibiotic stewardship across a large and diverse number of sites?
* How do determinants of implementation and needed strategies vary by context?
* What is the utility of a higher-resource implementation effort (named "Boost) focusing on outlier sites?

Data will be collected on number of children reached, adherence changes over time, types of implementation strategies employed, and characteristics of sites, prescribers, and patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months through 17 years
* ARTI diagnosis (acute otitis media (AOM), Group A Streptococcal (GAS) pharyngitis, acute sinusitis, and community-acquired pneumonia (CAP))

Exclusion Criteria:

* Age <6months or >18 years
* No ARTI diagnosis

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children meeting eligibility criteria and treated at any facility within the Intermountain region specified (wave 1 & wave 2) between January 1, 2026 and December 31, 2028.
Sampling Method: Non-Probability Sample
Enrollment: 259000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Guideline-adherent Broad vs. Narrow Spectrum Antibiotic Prescribing | Baseline month adherence and post implementation (12 months). Maintenance period is 6 months post implementation.
  Rates of narrow-spectrum antibiotic (AB) prescriptions as a proportion of all antibiotics prescribed in aggregate and within each of these diagnoses: Acute otitis media, Group A streptococcal pharyngitis, Acute sinusitis, and Pneumonia.
Guideline-adherent Duration of Antimicrobial Therapy | Baseline month adherence and post implementation (12 months). Maintenance period is 6 months post implementation.
  Rate of AB prescriptions with guideline-adherent number of days prescribed as proportion of all AB prescriptions in aggregate and for each of the target ARTI diagnoses.

SECONDARY OUTCOMES:
Rate of Treatment Failure | Baseline month adherence and post implementation (12 months). Maintenance period is 6 months post implementation
  Clinical encounter for the same diagnosis between 2 and 14 days following the index encounter and receipt of an alternative antibiotic for the same respiratory diagnosis during the return visit.
Adoption (Staff): Adherence to Protocols | Baseline month adherence and post implementation (12 months). Maintenance period is 6 months post implementation
  Number and proportion of prescribers who are "adherent" to guideline-based prescribing protocols for Broad vs. Narrow Spectrum AB Prescribing, and Duration.
Adoption (Organization): Adherence to Protocols | Baseline month adherence and post implementation (12 months). Maintenance period is 6 months post implementation.
  Number and proportion of sites where 60% of prescribers are adherent.

IPD SHARING:
Plan to Share IPD: No
This is an implementation study using observational data with a waiver of consent. Therefore, there is no consent to allow for the sharing of IPD.